CLINICAL TRIAL: NCT01915017
Title: Interventions to Improve Functional Outcome and Persistent Symptoms in Schizophrenia
Acronym: Mcog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Dawn Velligan, Professor, Director Division of Schizophrenia and Related Disorders, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH082793-03 (NIH)
Record Dates: First submitted 2013-07-26; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognitive Adaptation Training; Cognitive Behavior Therapy for Psychosis; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cognitive Behavior Therapy for Psychosis (Experimental): Cognitive behavior therapy for psychosis is a manual-driven collaborative talk-therapy designed to help the individual identify appraisal biases and cognitive distortion, identify alternative explanations for events, and find ways to cope with the distress caused by persistent psychotic symptoms.
  Interventions: Behavioral: Cognitive Behavior Therapy for Psychosis
- Cognitive Adaptation Training (Experimental): CAT is a manual driven treatment using environmental supports such as signs, alarms, checklists, electronic devices, and the organization of belongings to bypass cognitive and motivational impairments and to cue and sequence adaptive behavior.
  Interventions: Behavioral: Cognitive Adaptation Training
- Multi-modal Cognitive Therapy (Experimental): Combines Cognitive Behavior Therapy for Psychosis and Cognitive Adaptation Training into one home-delivered intervention
  Interventions: Behavioral: Multi-modal Cognitive Therapy
- Treatment as Usual (Active Comparator): Medication follow up and limited case management provided by the local community mental health center
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Psychosis — The CBT manual to be used for the present study was based upon the work of Kingdon and Turkington (2005) and Granholm et al., (2005) a group-delivered CBT skills training). Available manuals were modified to improve ease of training and to better accommodate the delivery of the full CBT treatment in the home environment. Supervision will be provided throughout the study by D. Turkington and S. Tai world renowned experts in CBT for psychosis. Training will be held for 1-2 weeks annually and supervision will proceed weekly via SKYPE. All therapists will be certified prior to providing treatment for the trial. Sessions are conducted weekly by master's and doctoral level therapists.
  Arms: Cognitive Behavior Therapy for Psychosis
Behavioral: Cognitive Adaptation Training — CAT supports are established and maintained on weekly home visits by bachelor's and master's level staff. Regular supervision will be provided by the PI who developed CAT.
  Arms: Cognitive Adaptation Training
Behavioral: Multi-modal Cognitive Therapy — A manual driven intervention combining CBT and CAT. Weekly sessions delivered in the home focus on altering cognitive biases using CBT and bypassing cognitive deficits using environmental supports
  Arms: Multi-modal Cognitive Therapy
Other: Treatment as Usual — Standard medication follow up and limited case management
  Arms: Treatment as Usual

SUMMARY:
Many individuals with schizophrenia continue to hear voices, have false beliefs, and problems with attention, memory planning and everyday functioning even with medication treatment. The process of recovery in schizophrenia involves treating the whole person. This study will test a new Multimodal Cognitive Treatment (Mcog). Mcog works around problems in attention, memory and planning by using supports in the home such as signs, checklists, and alarms to improve everyday functioning. Mcog also helps the individual to examine the evidence for their beliefs and to deal with symptoms like voices that are not completely resolved with medications. We will compare 4 treatments to determine if this combined approach improves both symptoms and functioning for individuals with schizophrenia.

DETAILED DESCRIPTION:
The process of recovery in schizophrenia involves resolving persistent symptoms and improving functional outcomes. Our research groups have demonstrated that using environmental supports in the patient's home to bypass deficits in cognitive functioning in a treatment called Cognitive Adaptation Training (CAT) improves adherence to medications and functional outcomes in schizophrenia and that Cognitive Behavior Therapy (CBT) decreases symptomatology and the negative effect of persisting symptoms upon individuals with this disorder. Data suggest these treatments have modality specific effects. Targeting both functional outcomes and persistent positive symptoms in a multimodal cognitive treatment provided in the patient's home is likely to have the most robust effects on functional outcomes, persistent symptoms and the distress caused by these symptoms for individuals with schizophrenia. We propose to randomize 200 individuals with schizophrenia taking antipsychotic medications to one of four psychosocial treatments for a period of 9 months: 1) CAT, 2) CBT, 3) Multimodal Cognitive Treatment (Mcog; an integrated treatment featuring aspects of both CAT and CBT), and 4) standard treatment as usual (TAU). Patients will be followed for 6 months after treatment is completed. Outcomes will be assessed at baseline and every 3 months. Primary outcome variables with include measures of symptomatology and functional outcome. We hypothesize that patients in treatments with CBT as a component (CBT and Mcog) will improve to a greater extent on measures of symptomatology than those randomized to non-CBT treatments (CAT or TAU)and that patients in Mcog will improve to a greater extent than those in single modality CAT. Moreover, we hypothesize that patients in treatments with CAT as a component (CAT and Mcog) will improve to a greater extent on measures of symptomatology than those randomized to non-CAT treatments (CBT or TAU) and that patients in Mcog will improve to a greater extent than those in single modality CAT. The potential public health implications of promoting recovery in schizophrenia through multi-modal treatments are profound. By integrating effective treatments the potential for synergistic improvement scan be assessed. Home visits can be costly. Maximizing the benefits to patients by providing multi-modal treatment on the same home visit is likely to improve a broader range of outcomes with minimal additional cost.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who have given informed consent.
2. Between the ages of 18 and 60.
3. Diagnosis of schizophrenia or schizoaffective disorder according to DSM-IV criteria as determined on the basis of the Structured Clinical Interview for Diagnosis Checklist (SCID-P) Checklist.
4. Receiving treatment with an oral atypical antipsychotic medication other than clozapine
5. Able to provide evidence of a stable living environment (individual apartment, family home, board and care facility) with no plans to move in the next year.
6. Intact visual and auditory ability as determined by a computerized screening battery.
7. Ability to read at the 5th grade level or higher based upon WRAT score.
8. Able to understand and complete rating scales and neuropsychological testing.
9. Delusions or hallucinations at a level of Moderate according to the BPRS. (Score of 4 or higher on items assessing hallucinations, unusual thought content, or suspiciousness.

Exclusion Criteria:

1. History of significant head trauma, seizure disorder, or mental retardation.
2. SOFAS scores >70 indicating a high level of social and occupational functioning.
3. Alcohol or drug abuse or dependence within the past 3 months.
4. Currently being treated by an ACT team.
5. History of violence in the past one year period.
6. Exposure to CAT treatment in that past 2 years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2008-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in Brief Psychiatric Rating Scale Psychosis Factor Score | baseline to 9 months
  Combines scores on BPRS for hallucinations, unusual thought content, suspiciousness and conceptual disorganization. Mean score varies from 1-7 with higher scores indicating more severe symptomatology
Change in Multnomah Community Ability Scale | Baseline to 9 months
  17-item scale assessing a variety of domains of community adjustment including Interference with functioning, Adjustment to living, Social competence, and Behavioral Problems. Higher scores reflect better community functioning.

SECONDARY OUTCOMES:
Change in Auditory Hallucination Rating Scale | Baseline to 9 months
  Examines the degree to which hallucinatory experiences are negative, distressing and disrupt the activities of the individual. The scale above separates how frequently the voices are distressing vs. non-distressing, the intensity of distress when the voices are distressing, the loudness of the voices and the degree of disruption in daily activities in separate items.
Change in Delusion Rating Scale | Baseline to 9 months
  Delusional ideas are rated with respect to the degree of conviction, the amount and duration of preoccupation, the amount and the level of distress experienced and the level of interference with activities.

OTHER OUTCOMES:
Change in Scale to Assess Unawareness of Mental Disorders | Baseline to 9 months
  Assesses insight into the illness, specific symptoms and the need for treatment.